CLINICAL TRIAL: NCT05425264
Title: Home-Based Exercise Tele-Rehabilitation in High-Risk Veterans: Impact of COVID-19 Exposure and Socioeconomic Factors
Brief Title: Home-Based Exercise Tele-Rehabilitation After COVID-19
Acronym: BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency); Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F3639-R
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Post SARS-CoV2 (COVID-19)
Keywords: Exercise; COVID-19; Cardiopulmonary
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Intervention Model Description: Exercise tele-rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tele-exercise (Experimental): Exercise training 2x/week at home. Sessions include circuit exercises of aerobic and resistive training stations which are led remotely.
  Interventions: Other: Tele-exercise

INTERVENTIONS:
Other: Tele-exercise — Exercise training 2x/week at home. Sessions include circuit exercises of aerobic and resistive training stations which are led remotely.

SUMMARY:
The Coronavirus Disease 2019 (COVID-19) pandemic has resulted in catastrophic infections and fatalities across the nation. Many older Veterans with comorbidities are especially vulnerable to complications and poor recovery. This award will investigate the effect of a novel, home-based, supervised, group exercise tele-rehabilitation in Veterans recovered from COVID-19 on cardiopulmonary and physical function.

DETAILED DESCRIPTION:
There is an urgent need to understand the lasting impact of COVID-19 on the cardiopulmonary system to improve physical function and prevent long-lasting disability. Pertinent knowledge gaps regarding the post-recovery physiology driving any impairments need to be addressed to improve the quality of life in Veterans with prior SARS-CoV-2 infection. Further, it is important to devise successful rehabilitation strategies that can be safely conducted in a Veteran's home. Hence, the investigators propose to utilize VA Video Connect to deliver a home based, supervised group exercise program to Veteran COVID-19 survivors. The objective of this exercise trial is to determine the influence of COVID-19 on cardiorespiratory fitness, pulmonary and physical function and to investigate the effect of a home-based exercise tele-rehabilitation on these outcomes. The study design includes rural and urban sites and investigators with a history of VA rehabilitation collaboration. Moreover, the investigators will explore healthcare disparities related to COVID-19 which are associated with functional decline and may affect sustainability of exercise rehabilitation strategies deployed, if necessary, under social distancing restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* documented COVID-19 > 90 days ago
* diagnosis of 2 of following conditions: hypertension, diabetes, cardiovascular disease, chronic kidney disease, chronic obstructive pulmonary disease OR 1 condition and BMI > 30 kg/m2

Exclusion Criteria:

* myocardial infarction (within 3 months)
* exertional or unstable angina (chest pain that limits activity)
* severe congestive heart failure (EF < 20% in last year or NYHA Classification III or IV)
* uncontrolled hypertension (SBP >180 &/or DBP > 110 mm Hg at screening)
* screening EKG with ischemia, complex arrhythmia, or high-grade block (per Minnesota Code)
* poorly controlled diabetes mellitus (FBS>200 mg/dl, RBS > 299 mg/dl, or HbA1C > 10)
* treatment for cancer except skin cancer (within 3 months)
* peripheral vascular disease with claudication
* severe arthritis limiting ambulation
* neurologic disease limiting ambulation (weakness requiring assist device; severe neuropathy)
* end stage liver disease (decompensated liver disease)
* End stage renal failure (dialysis)
* severe pulmonary disease (home O2, admission for dyspnea or pneumonia within 1 month)
* high fall risk (history of falls, bone fracture)
* dementia (based on Evaluation to Consent)
* signs or symptoms of any medical comorbidity that would preclude exercise testing or training
* exercises on routine basis (structured aerobic exercise > 3 time per week)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in VO2peak | Baseline and after 12 weeks tele-exercise
  physical fitness, units are ml/kg/min

SECONDARY OUTCOMES:
Change in 2-minute step test | Baseline and after 12 weeks tele-exercise
  physical function, units are number of times
chair stands | Baseline and after 12 weeks tele-exercise
  muscular strength, units are number of times

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No